CLINICAL TRIAL: NCT05513014
Title: Impact of Secukinumab on Clinical and Patient Reported Outcomes in Patients With Psoriasis in a Real World Setting in the US (Bionaive Secukinumab Users NVS 521)
Brief Title: Impact of Secukinumab on Clinical and Patient Reported Outcomes in Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457AUS31
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Secukinumab: Overall Cohort: Patients with Psoriasis who initiated Secukinumab
  Interventions: Drug: Secukinumab
- Biologic Experienced: Patients who had the history of use of ≥1 biologic medication for the treatment of PsO at the time of SEC initiation
- Biologic Naive: Patients who had no history of use of biologic medication for the treatment of PsO at the time of SEC initiation

INTERVENTIONS:
Drug: Secukinumab — Patients with Psoriasis who initiated Secukinumab
  Groups: Secukinumab: Overall Cohort

SUMMARY:
The study was conducted to describe the demographics, disease characteristics, disease severity, comorbidities and patient reported outcomes at baseline and follow-up periods among adult patients diagnosed with PsO in CorEvitas' PsO Registry under routine medical care initiating secukinumab (SEC).

DETAILED DESCRIPTION:
This is a retrospective analysis of a prospective observational cohort using CorEvitas' PsO registry of adult PsO patients. This study describes clinical and patient reported outcomes among adult patients initiating Secukinumab (SEC). Biologic experienced and naïve patients are examined separately. This study also describes changes in clinical and patient reported outcomes over time.

CorEvitas' Psoriasis Registry is a prospective, observational cohort of adult PsO patients starting systemic therapy, launched in April 2015 with sites in the US and Canada. Data collection occurs every ~6 months at routine dermatology visits. This study included US PsO patients who initiated secukinumab at or after enrollment and had a subsequent 6- and/or 12-month follow-up visit (Apr 2015 to Dec 2020).The index date is defined as the date of the first SEC initiation at or after enrollment.

ELIGIBILITY:
Inclusion Criteria:

The patient must:

* Have been diagnosed with PsO by a dermatologist.
* Be at least 18 years of age.
* Be willing and able to provide written informed consent for participation in the registry.
* Have started on or switched to an eligible systemic PsO treatment at enrollment1 or within the previous 12 months of the date of enrollment.

Exclusion Criteria:

* Patient is participating in or planning to participate in an interventional clinical trial with a nonmarketed or marketed investigational drug (i.e. phase I-IV drug trial).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with psoriasis who initiated Secukinumab
Sampling Method: Non-Probability Sample
Enrollment: 1518 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Age | Baseline
  Age was reported to describe the sociodemographic characteristics of the patients.
Gender | Baseline
  Gender was reported to describe the sociodemographic characteristics of the patients.
Race | Baseline
  Race was reported to describe the sociodemographic characteristics of the patients.
Ethnicity | Baseline
  Ethnicity was reported to describe the sociodemographic characteristics of the patients.
Body weight | Baseline
  Body weight was reported to describe the sociodemographic characteristics of the patients.
Number of patients: Weight category | Baseline
  Number of patients with Weight category were reported to describe the sociodemographic characteristics of the patients.
Number of patients: CDC BMI categories | Baseline
  Number of patients with CDC BMI categories were reported to describe the sociodemographic characteristics of the patients.
Number of patients: Smoking history | Baseline
  Number of patients with Smoking history were reported to describe the sociodemographic characteristics of the patients.
Number of patients: Alcohol use history | Baseline
  Number of patients with Alcohol use history were reported to describe the sociodemographic characteristics of the patients.
Number of patients: Insurance type | Baseline
  Number of patients with Insurance type were reported to describe the sociodemographic characteristics of the patients.
Number of patients: Provider region (US Census Bureau) | Baseline
  Number of patients with Provider region (US Census Bureau) were reported to describe the sociodemographic characteristics of the patients.
Psoriasis duration | Baseline
  Psoriasis duration was reported to describe the Disease characteristics of the patients.
Age at onset of PsO symptoms | Baseline
  Age at onset of PsO symptoms was reported to describe the Disease characteristics of the patients.
Number of patients: Morphology | Baseline
  Number of patients with Morphology were reported to describe the disease characteristics of the patients.
Number of patients: Comorbid psoriatic arthritis (PsA) | Baseline
  Number of patients with Comorbid psoriatic arthritis (PsA) were reported to describe the disease characteristics of the patients.
Psoriatic arthritis duration | Baseline
  Psoriatic arthritis duration was reported to describe the Disease characteristics of the patients.
Number of patients: History of comorbidities/toxicities | Baseline
  Number of patients with History of comorbidities/toxicities were reported to describe the disease characteristics of the patients.
Number of patients: History of IBD | Baseline
  Number of patients with History of IBD were reported to describe the disease characteristics of the patients.
Number of patients: Any infection | Baseline
  Number of patients with any infection were reported to describe the disease characteristics of the patients.
Dermatology Life Quality Index (DLQI) (Score: 0-30) | Baseline
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Number of patients: DLQI: Effect on life | Baseline
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Patient global assessment (PGA) | Baseline
  The PGA scoring system is based on response to treatment as measured by lesion erythema, induration, and scale, with score assignments that range from clear, almost clear, mild, moderate, to severe.
Patient itch assessment (VAS: 0-100) | Baseline
  Patient itch assessment was reported to evaluate overall, how severe was the itch from psoriasis in the past week. The score ranged from 0 to 100, where negative change indicated that the score declined over time.
Patient fatigue assessment (VAS: 0-100) | Baseline
  Patient fatigue assessment was reported to evaluate overall, how severe was the fatigue from psoriasis in the past week. The score ranged from 0 to 100, where negative change indicated that the score declined over time.
Patient skin pain assessment (VAS: 0-100) | Baseline
  Patient skin pain assessment was reported to evaluate overall, how severe was the skin pain from psoriasis in the past week. The score ranged from 0 to 100, where negative change indicated that the score declined over time.
Patient health state today (EQ-5D VAS: 0-100) | Baseline
  Questions: Given questions in the following 5 dimensions: (a) mobility, (b) self-care, (c) usual activities, (d) pain/discomfort and (e) anxiety/depression.
  With each dimension scored in 3 levels: 1 = {(a)-(c) =No problems, (d)=No pain, (e)=Not anxious or depressed}; 2 = {(a)-(c) = Some problems, (d) = Moderate pain or discomfort, (e ) = Moderately anxious or depressed}; 3={(a) = Confined to bed, (b)-(c)= Unable to do, (d) = Extreme pain or discomfort, (e) = Extremely anxious or depressed} With each dimension scored in 5 levels: 1 = No problems, 2 = Slight problems, 3 = Moderate problems, 4 = Severe problems, 5 = Extreme problems.
Number of patients: Mobility problems | Baseline
  Included the following: No problems, some problems, confined to bed
Number of patients: Self-care problems | Baseline
  Included the following: No problems, some problems, unable
Number of patients: Usual activities problems | Baseline
  Included the following: No problems
Number of patients: Some problems | Baseline
  Included the following: Unable
Number of patients: Pain or discomfort | Baseline
  Included the following: None, moderate and extreme
Number of patients: Work Productivity and Activity Impairment Questionnaire (WPAI) (0 to 100%) | Baseline
  Questions:1 = Currently employed? 2 = Hours missed due to psoriasis? 3 = Hours missed other reasons? 4 = Hours actually worked? 5 = Degree problem affected productivity while working (VAS (0 to 100) measurement)? 6 = Degree problem affected regular activities (VAS (0 to 100) measurement)? Scores: Multiply scores by 100 to express in percentages for reported categories: Percent work time missed due to problem: Q2/(Q2+Q4) Percent impairment while working due to problem: Q5/10 Percent overall work impairment due to problem: Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4)))x(Q5/10)] Percent activity impairment due to problem: Q6/10
PASI (Score: 0-72) | Baseline
  PASI (Score: 0-72) was reported to describe the PsO Specific Measures of the patients.
BSA (% involvement) | Baseline
  BSA (% involvement) was reported to describe the PsO Specific Measures of the patients.
Number of patients: BSA categorical | Baseline
  Number of patients with BSA categorical were reported to describe the PsO Specific Measures of the patients.
Number of patients: Investigator Global Assessment | Baseline
  Number of patients with Investigator Global Assessment were reported to describe the PsO Specific Measures of the patients.
Number of patients: PEST Score | Baseline
  Number of patients with PEST Score were reported to describe the PsO Specific Measures of the patients.
Number of patients: Therapies - Prior and Concomitant Drugs | Baseline
  Included the following:
  Unique prior biologic count Prior biologic exposures Unique prior non-biologic count Prior non-biologic exposures Nonbiologic naïve Current or prior topical use Concomitant non-biologic systemics
Number of patients: Primary reason for SEC initiation | Baseline
  Number of patients with Primary reason for SEC initiation

SECONDARY OUTCOMES:
Change from baseline in Investigator Global Assessment (IGA) | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
Change from baseline in PASI (Score: 0-72) | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
Change from baseline in BSA (% involvement) | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
Change from baseline in Patient health state today (EQ-5D VAS: 0-100) | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
Change from baseline in WPAI summary scores | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
Change from baseline in DLQI (Score: 0-30) | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
  The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Change from baseline in Patient global assessment | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
  The PGA scoring system is based on response to treatment as measured by lesion erythema, induration, and scale, with score assignments that range from clear, almost clear, mild, moderate, to severe.
Change from baseline in Patient itch assessment (VAS: 0-100) | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
  Patient itch assessment was reported to evaluate overall, how severe was the itch from psoriasis in the past week. The score ranged from 0 to 100, where negative change indicated that the score declined over time.
Change from baseline in Patient fatigue assessment (VAS: 0-100) | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
  Patient fatigue assessment was reported to evaluate overall, how severe was the fatigue from psoriasis in the past week. The score ranged from 0 to 100, where negative change indicated that the score declined over time.
Change from baseline in Patient skin pain assessment (VAS: 0-100) | Baseline, 6 and 12 months follow-up visits post index ( The index date is defined as the date of the first SEC initiation at or after enrollment i.e. Apr 2015 to Dec 2020)
  Changes in continuous outcomes between baseline, 6 and 12 month follow-up visit among patients remaining on SEC at 6 and 12 months, by prior biologic use.
  Patient skin pain assessment was reported to evaluate overall, how severe was the skin pain from psoriasis in the past week. The score ranged from 0 to 100, where negative change indicated that the score declined over time.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CAIN457AUS31 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17969